CLINICAL TRIAL: NCT03897114
Title: Cocoa Intake for the Prevention of Gastrointestinal Problems in Athletes: Effects on Oxidative Stress, Inflammation, Microbiota and Sports Performance
Brief Title: Cocoa Intake for Health Promotion in Athletes
Acronym: INDYCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Mar Larrosa, Tenure Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AGL2016-77288-R
Record Dates: First submitted 2019-03-04; First posted 2019-04-01 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Healthy Subjects
Keywords: Nutritional Supplement; Cocoa; Prebiotic; Physical Exercise; Gut Microbiota
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled study
Who Masked: Participant, Investigator
Masking Description: Cocoa and maltodextrin (placebo) are provided in identical sachets which are identified just with the letters A and B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cocoa group (Experimental): The cocoa will be provided in sachets. The intervention will be carried out for 10 weeks. Cocoa is provided in a single daily dose of 5 g, which contains 83 mg of flavonoids per gram of cocoa (dose at which a prebiotic effect has been shown).
  Interventions: Dietary Supplement: Cocoa group
- Placebo group (Placebo Comparator): Maltodextrin will be supplied as a placebo, which will be provided in sachets. Athletes will take 5g of product per day.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Cocoa group — Athletes perform the same training program and they take 5 g of cocoa (83 mg of flavonoids per gram of cocoa) mixed with low-fat milk for 10 weeks.
  Arms: Cocoa group
Dietary Supplement: Placebo group — The athletes perform the same training program and they take for 10 weeks 5 g maltodextrin mixed with low-fat milk for 10 weeks
  Arms: Placebo group

SUMMARY:
Athletes consume an extra of nutritional supplements every day with the purpose of improving their athletic performance, sometimes without being aware of their health. Cocoa could be a good nutritional supplement for athletes without causing them adverse effects. One of the most common health concerns in athletes are gastrointestinal problems. The cause of these problems seem to be a compendium of physiological and mechanical causes that are altered due to nutritional factors. Currently, there is no assay in which a nutritional intervention study has been proposed over time of training, in order to improve the gastrointestinal problems associated with the performance of physical exercise.

DETAILED DESCRIPTION:
The objective of this project is to investigate the benefits of daily consumption of cocoa in endurance athletes in:

A) Gastrointestinal problems associated with exercise. B) Reinforcement of the gastrointestinal barrier. C) Parameters of inflammation and oxidative stress. D) Sports performance. E) Body composition

The starting hypothesis of this project is based on the fact that daily cocoa consumption could improve the gastrointestinal symptoms associated with resistance exercise. Cocoa decreases the symptoms associated with splenic hypovolemia and strengthens the gastrointestinal epithelial barrier increasing the presence of Lactobacillus spp. and Bifidobacterium spp. in the intestinal microbiota.

A randomized, blinded, parallel placebo controlled intervention study will be carried out in endurance athletes who train in the sports facilities of the European University of Madrid. The number of male athletes for the study will be 56 (28 in each experimental group), all of them aimed at competition with an age between 18 and 40 years and an aerobic power consumption of oxygen greater than or equal to 55 mL / kg / min). The calculation of the sample size has been made selecting with a significance level alpha = 0.05 and a power (beta) of 0.90 for a 2-tailed analysis, taking into account we want to detect a difference of at least 15% in the improvement of the gastrointestinal symptoms, that the standard detected deviation in the questionnaire to be used, in previous studies, is 1.5 points out of 9 and that the expected proportion of losses is 15%.

Before and after the intervention, the athletes will do a test in which we will measure their maximum aerobic capacity. This will be done in the facilities of Europea University of Madrid where there is available a rolling belt. Also, they will do a second test in which we will measure the time they spend running a kilometer at the maximum speed. Body composition will be evaluated by dual-energy X-ray absorptiometry (DEXA). Blood, urine and feces samples will be required before and after the physical tests. Blood and urine samples will be collected in the morning while the feces samples will be collected the day before. The biological samples will be frozen at -80ºC until analyses.

The intervention will be carried out for 10 weeks. Cocoa or placebo will be provide in a single daily intake of 5 g of cocoa containing 500 mg of flavanols (dose at which a prebiotic effect has been demonstrated) or 5 g of maltodextrin.

ELIGIBILITY:
Inclusion Criteria:

* Men.
* Age between 18 and 50 years
* Aerobic power of oxygen consumption greater than or equal to 55 mL / kg / min

Exclusion Criteria:

* Intake of antibiotics (3 months before the trial) or any chronical medication.
* Intake of probiotics, prebiotics or any type of food or ergogenic supplements.
* To be vegetarian or vegan
* Smoke.
* Have documented gastrointestinal diseases (ulcers, irritable bowel, ulcerative colitis, Crohn's disease, etc.).
* Previous gastrointestinal surgeries or any disease diagnosed at the time of inclusion in the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — High performance sportsmen
Enrollment: 56 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Measurement of fat mass | Fat mass will be analyzed at the beginning (baseline dose) and after 10 weeks of intervention
  Energy X-ray absorptiometry (DEXA ).

SECONDARY OUTCOMES:
Measurement of lean mass | Lean mass will be analyzed at the beginning (baseline dose) and after 10 weeks of intervention
  Energy X-ray absorptiometry (DEXA ).
Sport performance test. | Sport performance will be analyzed at the beginning (baseline dose) and after 10 weeks of intervention
  Assessment of maximal aerobic capacity.
Sport performance test 2. | Sport performance will be analyzed at the beginning (baseline dose) and after 10 weeks of intervention
  Measurement of the time that the sportsmen spend running one kilometer at the maximum speed.
Change in eating habits. | Lifestyle will be analyzed at the beginning (baseline dose) and after 10 weeks of intervention.
  Food Frequency Questionnaire.
Change in Gut Microbiota | Gut microbiota will be analyzed at the beginning (basiline dose) and after 10 weeks of intervention.
  Determination of Microbial diversity by 16S rRNA Sequencing.
Measurement of the parameters of inflammation. | Plasma cytokines will be analyzed at the beginning and at the end of the 10-week intervention.
  Cytokines will be measured in plasma (IL-6, IL-10, IL-1β).
Indicators of gastrointestinal barrier. | Plasmatic LPS will be analyzed at the beginning and at the end of the 10-week intervention.
  Determination of plasmatic lipopolysaccharide (LPS) levels as an indicator of bacterial translocation.
Modification from baseline of gastrointestinal symptoms at 10 weeks | The questionnaire for the evaluation of gastrointestinal symptoms will be given to the athletes at the beginning and at the end of the 10-week intervention.
  The evaluation of gastrointestinal symptoms will be carried out through following the questionnaire described by Pfeiffer et al. (2009).
Change from baseline of oxidative stress parameters . | Nitric oxide will be analyzed at the beginning and at the end of the 10-week intervention.
  Nitric oxide levels will be measured in plasma and urine.

CONTACTS AND LOCATIONS:
Overall Officials: María del Mar Larrosa Pérez, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Jose Ángel García Merino, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided